CLINICAL TRIAL: NCT06459362
Title: Serum Cystatin C for Early Detection of Acute Kidney Injury After Primary Percutaneous Coronary Intervention
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shrook S. Ahmed, Demonstrator, Assiut University
Other Study IDs: SSAS
Record Dates: First submitted 2024-05-31; First posted 2024-06-14 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Serum cystatin C — Diagnostic test for detection of acute kidney injury

SUMMARY:
This study aims to evaluate whether the serum levels of Cystatin C (CysC) can be used as early biomarkers for the identification of patients who are prone to AKI after cardiac interventional surgeries as primary percutaneous coronary intervention (PCI)

DETAILED DESCRIPTION:
Acute Kidney Injury (AKI) is defined as an absolute increase in serum creatinine ≥0.3 mg/dl (≥26.4 μmol/l), a percentage increase in serum creatinine ≥50% (1.5-fold from baseline), or a reduction in urine output (documented oliguria < 0.5 ml/kg/hour for > 6 hours) Serum creatinine which is considered the gold standard currently for diagnosis of AKI remains unchanged until 50% of kidney function falls down. It is affected by non-specific factors like diet, age, dehydration, muscle mass, gender, and drugs There were evidences of the association between AKI and acute coronary syndrome (ACS); First, AKI detection may be missed by cardiologists. Physicians tend to disregard mild or transient serum creatinine elevation during hospital stay for ACS, and they often attribute small serum creatinine increases to laboratory variations.

Cystatin C (CysC), a cystatin protease inhibitor, is less affected by non-specific factors. When GFR decreases, CysC begins to increase. CysC was recommended to be measured in addition to creatinine in GFR estimation.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Patient with absolute increase in serum creatinine ≥0.3 mg/dl (≥26.4 μmol/l) or with percentage increase in serum creatinine ≥50% (1.5-fold from baseline)
3. Patient with reduction in urine output (documented oliguria < 0.5 ml/kg/hour for > 6 hours)
4. Patient with typical chest pain, ECG changes, Echocardiogram positive finding

Exclusion Criteria:

1. History of nephrectomy
2. patient with renal transplantation
3. patient with renal replacement therapy initiated before admission
4. patient with chronic kidney disease
5. patient on regular haemodialysis
6. patient known to be diabetic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with typical chest pain and treated by primary percutaneous intervention
Sampling Method: Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
prevention and screening for early detection of acute kidney injury | 2 years
  using serum levels of Cystatin C (CysC) as early biomarkers for the identification of patients who are prone to AKI after cardiac inteventional surgeries as primary percutaneous coronary intervention (PCI)

IPD SHARING:
Plan to Share IPD: No